CLINICAL TRIAL: NCT04539392
Title: Assessment of the Sexuality of the Infertile Couple: Prospective Cohort Study
Brief Title: Assessment of the Sexuality of the Infertile Couple
Acronym: INFEXO
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2019-2/SH-01
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infertile couple
  Interventions: Other: Questionnaires on sexuality

INTERVENTIONS:
Other: Questionnaires on sexuality — Panel of questionnaires assessing sexuality, relationship satisfaction, and body image

SUMMARY:
The study hypothesis is that infertile couples experience an impact of their sexuality impacted during the diagnostic process carried out as part of the medically assisted procreation assessment, and also by the announcement of the possible cause of the couple's infertility. It is also conceivable that a disorder of the couple's sexuality forms the origin of, or is a contributor to, infertility.

ELIGIBILITY:
Inclusion Criteria:

* Couple in which each of the two partners has signed the consent form which is presented separately and independently of their partner.
* The patient must be a member or beneficiary of a health insurance plan
* Heterosexual infertile couple (according to the WHO definition) monitored at the Nîmes University Hospital in the urology / gynecology departments.

Adult patient (≥18 years old) and under 43 years old for women, 60 years old for men

Exclusion Criteria:

* The subject is participating in a category 1 interventional study, or is in a period of exclusion determined by a previous study
* One member of the couple refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient without good level of written and spoken French

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 80 heterosexual infertile couples (according to the WHO definition) followed at the Nîmes University Hospital in the Urology / Gynecology departments.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Sexuality of the female of the couple | 2 weeks after inclusion (start of MAP)
  Female sexual function index: The total score is between 2 and 36 with sexual dysfunction indicated for scores below 26.55
Sexuality of the female of the couple | 1 month after ovarian ponction (end of MAP)
  Female sexual function index: The total score is between 2 and 36 with sexual dysfunction indicated for scores below 26.55
Sexuality of the male of the couple | 2 weeks after inclusion (start of MAP)
  Male Sexual Health Questionnaire
Sexuality of the male of the couple | 1 month after ovarian ponction (end of MAP)
  Male Sexual Health Questionnaire
Ejactulation of the male of the couple | 2 weeks after inclusion (start of MAP)
  Premature Ejaculation Profile
Ejactulation of the male of the couple | 1 month after ovarian ponction (end of MAP)
  Premature Ejaculation Profile

SECONDARY OUTCOMES:
Sexuality of the female of the couple | 1 month after ovarian ponction (end of MAP)
  Female sexual function index: The total score is between 2 and 36 with sexual dysfunction indicated for scores below 26.55
Sexuality of the male of the couple | 1 month after ovarian ponction (end of MAP)
  Male Sexual Health Questionnaire
Body satisfaction and global self-perception of both members of the couple | 2 weeks after inclusion (start of MAP)
  Questionnaire de satisfaction corporelle et de perception globale de soi (QSCPGS): total score ranges from -100 to +100.
Body satisfaction and global self-perception of both members of the couple | 1 month after ovarian ponction (end of MAP)
  Questionnaire de satisfaction corporelle et de perception globale de soi (QSCPGS): total score ranges from -100 to +100.
Relationship satisfaction of both members of the couple | 2 weeks after inclusion (start of MAP)
  Dyadic Adjustment Scale-16 Distress if score less than 92 and without distress if the score is higher than 107
Relationship satisfaction of both members of the couple | 1 month after ovarian ponction (end of MAP)
  Dyadic Adjustment Scale-16 Distress if score less than 92 and without distress if the score is higher than 107
Self-esteem of both members of the couple | 2 weeks after inclusion (start of MAP)
  Rosenberg self-esteem scale: The score is between 10 and 40. A score below 25 indicates very low self-esteem. A score between 25 and 31 indicates low self-esteem. A score between 31 and 34 indicates average self-esteem. A score between 34 and 39 indicates strong self-esteem. A score above 39 indicates very high self-esteem.
Self-esteem of both members of the couple | 1 month after ovarian ponction (end of MAP)
  Rosenberg self-esteem scale: The score is between 10 and 40. A score below 25 indicates very low self-esteem. A score between 25 and 31 indicates low self-esteem. A score between 31 and 34 indicates average self-esteem. A score between 34 and 39 indicates strong self-esteem. A score above 39 indicates very high self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Huberlant, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France